CLINICAL TRIAL: NCT02352064
Title: EVALUATION OF THE DIAGNOSTIC VALUE OF PET (18F-FDG) IN CHRONIC GRAFT VERSUS HOST DISEASE (cGVH)
Acronym: TEP-GVH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00724-43
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET-CT at day 150+/-15 days (Experimental): Patient will have PET (18-FDG) following allogeneic stem cell transplantation
  Interventions: Procedure: PET (18-FDG)

INTERVENTIONS:
Procedure: PET (18-FDG) — Every patient will have a PET

SUMMARY:
Allogeneic stem cell transplantation was developed to cure many patients with hematological malignancies. It results in the development of graft versus host disease (GVHD) in 30-70% of cases. Chronic GVHD diagnosis currently uses biopsies of affected organs (skin, liver, gastrointestinal tract) and / or the observation of typical clinical signs sufficient for diagnosis. However, the anatomical sites for biopsy including the digestive tract are not clearly identified (high or low biopsy) and may present risks in their realization in particular in patients weakened by blood disease or immunosuppression.

PET-CT with 18F-FDG has already been evaluated in chronic inflammatory diseases such as Crohns disease with good sensitivity and specificity. It interest in the graft against the host was studied in acute forms of digestive and allows lesion mapping and monitoring the effectiveness of treatment.

Among patients with chronic GVHD scleroderma form, PET with 18F-FDG enabled to view musculoskeletal uptakes localized to the affected areas identified with MRI.

The investigators propose a study evaluating the sensitivity and specificity of the examination by PET-CT with 18F-FDG in the diagnosis of chronic GVHD compared to conventional diagnostic tools.

DETAILED DESCRIPTION:
Patients will have PET/CT at day 150+/-15d post-hematopoietic stem cell transplantation (HSCT)

ELIGIBILITY:
Inclusion Criteria:

* adult >18 years
* Signed informed consent
* subject covered by a social security system
* Absence of contraindication to PET (18F-FDG)
* Allogeneic stem cell transplantation

Exclusion Criteria:

* Adult patient under tutelage.
* Pregnant or lactating women or women of childbearing potential not currently practicing an adequate method of contraception
* Age<18 years
* Evolutive infectious disease
* glycemia >10mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Measure of sensibility and specificity of PET (18F-FDG) for cGVH diagnosis in comparison to standard care | 5 months
  Presence of pathological 18-FDG uptakes on PET-CT examination in allografted patient compared with standard tests (clinical examination score GVHD, as defined by the NI (with or without targeted organ biopsy) Patient with negative PET-CT and without GVHD signs (NIH classification according to Filipovitch et al) are considered as true negative. Patient with positive PET-CT without GVHD signs are considered as false positive. Patient with clinical GVHD and negative PET-CT are considered as falsse negative and patients with clinical GVHD and positive PET-CT are true positive. The follow-up will determine if PET-CT is positive before the onset of clinical signs of GVHD.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France